CLINICAL TRIAL: NCT03089086
Title: South Australian Meningococcal B Vaccine Herd Immunity Study
Acronym: B Part of It
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: SA Health (Other)
Responsible Party: Principal Investigator, Helen Marshall, Director, Vaccinology and Immunology Research Trials Unit, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HREC/16/WCHN/140; ACTRN12617000079347 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Meningococcal Disease
Keywords: meningococcal B vaccine; herd immunity; adolescents; young adults; south australia
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: A cluster randomised controlled trial to assess the impact of meningococcal B vaccine 4CMenB on nasopharyngeal carriage of N. Meningitidis
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Students within schools randomised to group A will receive two doses of licensed 4CMenB vaccine after baseline oropharyngeal swab with an interval of 1 to 2 months between doses, with the first dose given at the baseline visit in 2017.
  Interventions: Biological: Licensed 4CMenB vaccine
- Group B (No Intervention): Students within schools randomised to group B will receive the licensed 4CMenB vaccine following completion of baseline and 12 month oropharyngeal swab in 2018.

INTERVENTIONS:
Biological: Licensed 4CMenB vaccine — Two doses (0.5 mL each) of Bexsero ® vaccine at least 1 month to <3 months apart in adolescents.
  Other Names: Bexsero®
  Arms: Group A

SUMMARY:
To estimate the effect on carriage, all year 10, 11, and 12 students will be offered 4CMenB vaccination in South Australia through schools over the study period with 50% of the students enrolled receiving the vaccine in 2017 and 50% in 2018. In year 10 and 11 students, posterior pharyngeal swabs will be obtained at baseline and 12 months post baseline to estimate the difference in carriage prevalence of all genogroups of N. meningitidis between vaccinated and unvaccinated participants.

DETAILED DESCRIPTION:
This cluster randomised controlled study will be conducted in the context of funded 4CMenB vaccine offered to all students in years 10, 11, and 12.

Year 10 and 11 students will undergo baseline and 12 months posterior pharyngeal swabs. Year 12 students will undergo baseline posterior pharyngeal swabs only.

Randomisation will take place at the school level and will be stratified by school size ((<60, 60 to 119, and ≥120 students per year level) and school socio-economic status (SES), as measured by the Index of Community Socio-Educational Advantage (ICSEA); (ICSEA <970, 970 to 1020, >1020) For the purposes of the study a school is defined as an educational institution at which students in years 10, 11, 12 physically attend school during the week. All 260 schools in metropolitan and rural SA will be approached to participate in the study. All schools agreeing to participate will be randomised to 4CMenB vaccine in 2017 or 2018. Students at schools randomised to receive the vaccine at baseline will receive the 4CMenB vaccine in 2017. Students at schools randomised to receive the vaccine at the 12 month posterior pharyngeal swab will receive the 4CMenB vaccine in 2018.

Primary Objectives

• Estimate the difference in carriage prevalence of disease causing genogroup of N. meningitidis (A, B, C, W, X, Y) following the 12 month pharyngeal swab in year 10 and 11 students who received two doses of Bexsero®, compared to unvaccinated students.

Secondary objectives

* Estimate the difference in carriage prevalence of each disease causing genogroup of N. meningitidis (A, B, C, W, X, Y) following the 12 month pharyngeal swab in year 10 and 11 students who received two doses of Bexsero®, compared to unvaccinated students.
* Estimate the difference in carriage prevalence of all genogroups of N. meningitidis following the 12 month pharyngeal swab in year 10 and 11 students who received two doses of Bexsero ®, compared to unvaccinated students.
* Estimate the difference in acquisition (negative at baseline, positive at 12 month followup) of carriage of disease causing genogroups of N. meningitidis (A, B, C, W, X, Y) over a 12 month period in students who received two doses of Bexsero ®, compared to unvaccinated students.
* Estimate the difference in acquisition (negative at baseline, positive at 12 month followup) of carriage of all genogroups of N. meningitidis over a 12 month period in students who received two doses of Bexsero ®, compared to unvaccinated students
* Identify characteristics associated with carriage prevalence of all genogroups N. meningitidis in South Australian school students at baseline and 12 months.
* Identify characteristics associated with carriage prevalence of disease causing genogroups of N. meningitidis (A, B, C, W, X, Y) in South Australian school students at baseline and 12 months.

Exploratory objectives

* Describe changes in invasive meningococcal rates (attack rates) across all age groups pre and post 4CMenB vaccine intervention in South Australia.
* Describe N. meningitidis carriage density in year 10, 11, and 12 students using qPCR at baseline and 12 months in both vaccinated and unvaccinated students.
* Describe genome sequencing of N. meningitidis disease causing (A, B, C, W, X, Y) sequence types in year 10, 11, and 12 students at baseline and at 12 months.
* In schools randomized to Group A, describe the association of carriage prevalence of disease causing genogroups and vaccine uptake at school level following implementation.
* In schools randomized to Group A, describe the association of carriage prevalence of all N. meningitidis and vaccine uptake at school level following implementation.

ELIGIBILITY:
Inclusion criteria:

* South Australian secondary school students in years 10, 11, and 12 in 2017
* Written parental consent for those under the age of 18
* Written student consent assent for those under the age of 18 (or if 18 years old and older consent for themselves)
* Available at school for at least the first pharyngeal swab and willing to comply with study procedures

Exclusion Criteria:

1. Previous anaphylaxis following any component of Bexsero vaccine
2. Previous receipt of meningococcal B vaccine (Bexsero)
3. Known pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34489 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of all disease causing genogroups of N. meningitidis (A, B, C, W, X, Y) | 12 months
  As measured by PCR at 12 months in vaccinated and unvaccinated year 10 and 11 school students

SECONDARY OUTCOMES:
Prevalence of each N. meningitidis genogroup (A, B, C, W, X, Y) | 12 months
  As measured by PCR at the 12 month pharyngeal swab in vaccinated and unvaccinated year 10 and 11 school students
Prevalence of all N. meningitidis genogroups | 12 months
  As measured by PCR at the 12 month pharyngeal swab in vaccinated and unvaccinated year 10 and 11 school students
Acquisition of disease causing N. meningitidis (A, B, C, W, X, Y) genogroups (negative at baseline, positive at 12 month followup) | 12 months
  As measured by PCR in vaccinated and unvaccinated year 10 and 11 school students
Acquisition of all N. meningitidis | 12 months
  As measured by PCR in vaccinated and unvaccinated year 10 and 11 school students
Risk factors associated with carriage prevalence of all N. meningitidis | Baseline and 12 months
  As measured by PCR at baseline and 12 months
Risk factors associated with carriage prevalence of disease causing N. meningitidis | Baseline and 12 months
  As measured by PCR at baseline and 12 months

OTHER OUTCOMES:
Age specific IMD attack rates | Prior to and following implementation of the intervention
  Age specific IMD attack rates (per 100,000 population) in all age groups in South Australia
Carriage density of N. meningitidis (all genogroups) | Baseline and 12 months
  as measured by qPCR in year 10, 11 and 12 school students at baseline and 12 months
Description of whole genome sequences of carriage isolates | Baseline and 12 months
  Description of whole genome sequences of isolates known to cause disease (serogroup B, W, Y, C)
Whole genogroup sequencing of all carriage isolates | Baseline and 12 months
  Description of whole genome sequences of isolates
Vaccine uptake and carriage prevalence of all N. meningitidis. | 12 months
  Carriage prevalence as measured by PCR
Vaccine uptake and carriage prevalence of disease causing N. meningitidis. | 12 months
  Carriage prevalence as measured by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Helen Marshall, Principal Investigator — University of Adelaide
Locations (1):
- Vaccinology & Immunology Research Trials Unit, North Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data underlying published results will be available.
Supporting Information: Study Protocol, SAP
Time Frame: We estimate the data will be available from the start of 2021 for approximately 12 months.
Access Criteria: IPD will be made available on a case-by-case basis at the discretion of the International Scientific Advisory Committee and WCHN HREC. IPD data will only be available to achieve the aims in the approved proposal.

REFERENCES:
- [Background] Marshall HS, McMillan M, Koehler A, Lawrence A, MacLennan JM, Maiden MCJ, Ramsay M, Ladhani SN, Trotter C, Borrow R, Finn A, Sullivan T, Richmond P, Kahler CM, Whelan J, Vadivelu K. B Part of It protocol: a cluster randomised controlled trial to assess the impact of 4CMenB vaccine on pharyngeal carriage of Neisseria meningitidis in adolescents. BMJ Open. 2018 Jul 10;8(7):e020988. doi: 10.1136/bmjopen-2017-020988. PMID 29991629
- [Derived] McMillan M, Wang B, Koehler AP, Sullivan TR, Marshall HS. Impact of Meningococcal B Vaccine on Invasive Meningococcal Disease in Adolescents. Clin Infect Dis. 2021 Jul 1;73(1):e233-e237. doi: 10.1093/cid/ciaa1636. PMID 33587122
- [Derived] Marshall HS, Koehler AP, Wang B, A'Houre M, Gold M, Quinn H, Crawford N, Pratt N, Sullivan TR, Macartney K. Safety of meningococcal B vaccine (4CMenB) in adolescents in Australia. Vaccine. 2020 Aug 18;38(37):5914-5922. doi: 10.1016/j.vaccine.2020.07.009. Epub 2020 Jul 22. PMID 32712083
- [Derived] McMillan M, Walters L, Sullivan T, Leong LEX, Turra M, Lawrence A, Koehler AP, Finn A, Andrews RM, Marshall HS. Impact of Meningococcal B (4CMenB) Vaccine on Pharyngeal Neisseria meningitidis Carriage Density and Persistence in Adolescents. Clin Infect Dis. 2021 Jul 1;73(1):e99-e106. doi: 10.1093/cid/ciaa610. PMID 32447370
- [Derived] Marshall HS, McMillan M, Koehler AP, Lawrence A, Sullivan TR, MacLennan JM, Maiden MCJ, Ladhani SN, Ramsay ME, Trotter C, Borrow R, Finn A, Kahler CM, Whelan J, Vadivelu K, Richmond P. Meningococcal B Vaccine and Meningococcal Carriage in Adolescents in Australia. N Engl J Med. 2020 Jan 23;382(4):318-327. doi: 10.1056/NEJMoa1900236. PMID 31971677